CLINICAL TRIAL: NCT04969458
Title: Reliability and Validity of the Turkish Version of the Graded Chronic Pain Scale 2.0
Brief Title: Reliability and Validity of the Turkish Version of the GCPS 2.0.(Graded Chronic Pain Scale 2.0)
Acronym: GCPS
Status: Completed | Type: Observational
Sponsor: Yeditepe University (Other)
Responsible Party: Sponsor
Other Study IDs: 123456789
Record Dates: First submitted 2021-07-13; First posted 2021-07-20 (Actual); Last update posted 2021-07-20 (Actual); Status verified 2021-07

CONDITIONS: Chronic Pain; Scale Reliability Validity
Keywords: Graded Chronic Pain Scale; Chronic Pain; Disability; Chronic Low Back Pain; Validity and Reliability
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- participants: The study included individuals whose native language is Turkish, who are over the age of 18 and under the age 70, diagnosed with chronic low back pain, without Psychiatric disorder, Cognitive impairment, Dementia, or Alzheimer's and who want to participate in the study.
  Interventions: Other: survey application

INTERVENTIONS:
Other: survey application — Data collection tools used in the study;
  * Clinic and Demographic Evaluation Form
  * Oswestry Low Back Pain Disability Index (ODI)
  * Patterns of Activity Measure Pain (POAM-P)
  * Roland-Morris Disability Questionnaire (RMDQ)
  * Hospital Anxiety and Depression Scale (HADS)
  * Graded Chronic Pain Scale Version 2.0 (GCPS 2.0)

SUMMARY:
This study was designed to conduct Turkish adaptation, cross-cultural adaptation, validity, and reliability study of Graded Chronic Pain Scale 2.0 in order to use it for Turkish people with Chronic Pain.

DETAILED DESCRIPTION:
The GCPS 2.0 is an eight-item scale that evaluates the severity of chronic pain, the presence of persistent pain due to pain days, and the degree of disability due to pain. It is easy, simple, useful and multidimensional. 80 volunteer participants who had chronic low back pain were studied.The data collection tools used in this study were; Clinic and Demographic Evaluation Form, Oswestry Low Back Pain Disability Index, Patterns of Activity Measure Pain, Roland-Morris Disability Questionnaire, Hospital Anxiety, and Depression Scale, and Graded Chronic Pain Scale 2.0. In this study, the forms were sent by e-mail. The Snowball sampling method was used in the data collection process.The stages of the Beaton Protocol were followed in the translation of the scale. Validity was evaluated with the Face, Content, and Construct validity analyses. Exploratory and confirmatory factor analyses were applied to determine the construct validity of the Turkish version of the scale. Reliability was evaluated with the test-retest method, the parallel forms method, and the internal consistency. Ten days after completing the scale, 30 participants filled out the scale again for the Test-retest method. One of the scales we used for the parallel forms method was RMDQ and the other was ODI.

ELIGIBILITY:
Inclusion Criteria:

Participants were Turkish speakers and volunteer participants aged 18 years and over and under 70 years of age who had recurrent or persistent chronic LBP for 6 months or more.The following participants with CLBP diagnosed by a physician were included in the study. These;

* Disc herniations
* Mechanical back pain
* Lumbar strain
* Spondylolisthesis
* Degenerative disc disease
* Muscle imbalance
* Lumbago
* A trigger point in the back muscles

Exclusion Criteria:

* Having a history of illness such as Psychiatric disorder, Cognitive impairment, Dementia, or Alzheimer's
* Low back pain that needs immediate treatment (neoplasm, cauda equina syndrome, infection, fracture)
* Inflammatory low back pain
* Low back pain due to a vascular cause

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult, Older Adult
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2020-10-22 (Actual); Primary Completion 2020-11-16 (Actual); Study Completion 2020-11-23 (Actual)

PRIMARY OUTCOMES:
Graded Chronic Pain Scale 2.0 | 3 minutes
  GCPS 2.0 measures multiple dimensions of pain in patients with chronic pain.
Clinic and Demographic Evaluation Form | 5 minutes
  n the clinical section, there are questions the inclusion and exclusion criteria. According to this section, the patient is included in the study. In the demographic section, there is the section where the patient's demographic variables are collected.
Oswestry Low Back Pain Disability Index (ODI) | 5 minutes
  ODI is a questionnaire measuring the effect of low back pain on daily life and the level of disability caused by this pain.
Roland-Morris Disability Questionnaire (RMDQ) | 5 minutes
  RMDQ is a sensitive tool that measures the loss of function and disability due to low back pain.

SECONDARY OUTCOMES:
Hospital Anxiety and Depression Scale (HADS) | 5 minutes
  The hospital anxiety and depression scale have two sub-scales: Anxiety and Depression. 7 single-digit questions in the scale measure anxiety, while 7 questions with two numbers measure depression.
Patterns of Activity Measure Pain (POAM-P) | 15 minutes
  Some established activity patterns reduce patients' quality of life with chronic pain, increase their pain, and limit their movement. These are modified patterns such as Overdoing, Avoidance, Pacing. POAM-P determines which of these patterns chronic pain patients use. There are 10 questions in each subsection, also 30 questions in total.

CONTACTS AND LOCATIONS:
Locations (1):
- Yeditepe University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No